CLINICAL TRIAL: NCT05013125
Title: Assessment of Efficacy of ENDO-AID Assisted Colonoscopy in Adenoma Detection: a Single Centre Randomised Controlled Trial
Brief Title: ENDO-AID Assisted Tandem Colonoscopy RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kaori Futaba, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CREC.2021.336
Record Dates: First submitted 2021-07-26; First posted 2021-08-19 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Neoplasms
Keywords: Computer aided Polyp detection; Colonoscopy; Polyp detection; Colorectal polyps; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Colonoscopy - ENDO-AID assisted Colonoscopy (No Intervention): Patients will undergo usual colonoscopy as per usual practice, followed back to back by ENDO-AID assisted colonoscopy
- ENDO-AID assisted Colonoscopy - ENDO-AID assisted Colonoscopy (Active Comparator): Patients will undergo ENDO-AID assisted colonoscopy with all polyps treated as per usual practice, followed back to back by ENDO-AID assisted colonoscopy
  Interventions: Diagnostic Test: ENDO-AID CADe assisted Colonoscopy

INTERVENTIONS:
Diagnostic Test: ENDO-AID CADe assisted Colonoscopy — ENDO-AID is a dedicated endoscopy Computer-Aided Diagnosis (CADe) system where suspicious lesions are automatically detected and highlighted on the main monitor in real-time, alerting the endoscopist during the procedure.
  Arms: ENDO-AID assisted Colonoscopy - ENDO-AID assisted Colonoscopy

SUMMARY:
This study hypothesizes that more adenomas will be detected using the ENDO-AID assisted Colonoscopy compared to conventional colonoscopy.

A single-centre, randomized, same-day, back-to-back tandem colonoscopy trial comparing Adenoma Missed Rate and Adenoma Detection Rate in ENDO-AID assisted colonoscopy and conventional colonoscopy.

DETAILED DESCRIPTION:
Colorectal cancer is the third common cancer in the world and the commonest cancer in Hong Kong. Most sporadic colorectal cancers arise from benign polyps via adenoma-carcinoma sequence or the serrated polyp-carcinoma sequence. There are reports of unexpectedly high risk of interval carcinomas, as high as up to 9%, raising concerns about the effectiveness of colonoscopy in preventing colorectal cancers. Different techniques have been described to improve the area of mucosa visualised but lesions may still be missed due to failure of identification by the endoscopist.

Computer Aided diagnosis (CAD) assisted colonoscopy is becoming increasingly popular to address human error. Deep learning technology has surpassed human learning and advancement in technology now allows real-time Artificial Intelligence to assist colonoscopists in polyp detection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18years or above
* Referred to endoscopy unit for diagnostic or surveillance colonoscopy

Exclusion Criteria:

* Familial history of Familial adenomatous polyposis / Hereditary non-polyposis colorectal cancer
* Known history of inflammatory bowel disease
* Known colitis or suspicion of colitis (inflammatory bowel disease, diverticulitis, infective colitis)
* Emergency endoscopy of any nature (eg gastrointestinal bleeding, colonic decompression)
* Previous incomplete colonoscopy (not including insufficient preparation) / difficult colonoscopy
* Patients referred for a therapeutic procedure or assessment of a known non-resected lesion
* Patients with known palliative colorectal malignancy
* Patient with coagulopathy
* Patient with colostomy
* Patient with multiple co-morbidities (American Society of Anaesthesiologist >3)
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Adenoma missed rate | End of study, about 1 year
  To compare the adenoma missed rate (AMR) between ENDO-AID assisted Colonoscopy and conventional colonoscopy. AMR is defined as the number of adenomas detected in the second pass colonoscopy divided by the total number of adenomas detected in both passes for the same patients.

SECONDARY OUTCOMES:
Polyp missed rate | End of study, about 1 year
  To compare the Polyp missed rate (PMR) between ENDO-AID assisted Colonoscopy and conventional colonoscopy. PMR is defined as the number of polyps detected in the second pass colonoscopy divided by the total number of polyps detected in both passes for the same patients.
Adenoma detection rate | End of study, about 1 year
  To compare the Adenoma detection rate (ADR) between ENDO-AID assisted Colonoscopy and conventional colonoscopy for the first pass colonoscopy. ADR is defined as the proportion of patients with at least 1 adenoma detected in the first pass colonoscopy.
Patient missed rate | End of study, about 1 year
  To compare the patient missed rate (PMR) between ENDO-AID assisted colonoscopy and conventional white light colonoscopy. PMR is defined as the number of patients in whom adenomas were detected for the first time during second pass colonoscopy divided by the number of patients with at least 1 adenoma detected.
Number of polyps removed | End of study, about 1 year
  To compare the number of polyps removed between ENDO-AID assisted Colonoscopy and conventional white light colonoscopy
Baseline Parameters | End of study, about 1 year
  Baseline Parameters will be compared, including withdrawal time and Boston Bowel Preparation Scale in the first colonoscopy procedures
Serious Adverse Events | At 30 days
  To compare the Serious Adverse Events between ENDO-AID assisted Colonoscopy and conventional white light colonoscopy
Number of CAD assisted abnormality | End of study, about 1 year
  Number of abnormalities highlighted on ENDO-AID and actual number of abnormalities found macroscopically and histologically

CONTACTS AND LOCATIONS:
Overall Officials: Kaori Futaba, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, Chinese University of Hong Kong, Shatin, New Territories, Hong Kong